CLINICAL TRIAL: NCT04544332
Title: The GAIN Study: Understanding What Helps Children Learn to Like and Eat New Foods
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Temple University (Other); Global Alliance for Improved Nutrition (Other); Purdue University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2308
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Food Preferences; Parenting
Keywords: Infant Feeding; Toddler Feeding; Food Acceptance; Food Parenting
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unsweetened Supplement: Infants will receive 10 exposures to the unsweetened small quantity lipid nutritional supplement (SQ-LNS) at home
- Sweetened Supplement: Infants will receive 10 exposures to the sweetened small quantity lipid nutritional supplement (SQ-LNS) at home

SUMMARY:
Nutrition supplements have tremendous impact upon the nutritional and developmental status of malnourished children. These products have been designed to be acceptable to children (often by adding nutritive sweeteners to make them more palatable), but to date there has been little rigorous testing of their palatability for infants, toddlers and young children. The overall goal of this project is to investigate whether:

1. children's acceptance of a nutrition supplement is associated with maternal persistence in offering the food to her child over a 2-week period;
2. an unsweetened version of the nutrition supplement differs in short- and long-term acceptance; and
3. maternal liking of the supplement is associated with her persistence in offering the food to her child.

DETAILED DESCRIPTION:
More rigorous pre-testing of nutrition supplements, with a focus on palatability (i.e., observations of behavioral and facial responses to its taste) and its relation to children's acceptance (defined here as consumption), could provide important insights into the capacity for these products to transition from being perceived as "medicine" to being accepted as "food," or part of the usual child diet. A clearer understanding of the relation between observed child indicators of palatability and acceptance, both initially and over time (i.e., repeated exposure effects), is important for predicting the longer-term impacts on children's dietary intake, growth and health. Further, a better grasp of caregiver perceptions of the acceptability of these products, both their child's and their own, is critical in paving the way for overcoming barriers and identifying facilitators associated with longer-term acceptance of these nutritional supplements.

We secondarily will also explore the effects of potential mediators on caregiver persistence and infant acceptance of a sweetened and an unsweetened small-quantity lipid nutrition supplement (SQ-LNS) such as:

* Maternal feeding self-efficacy
* Caregiver food neophobia
* Caregiver feeding styles using the Infant Feeding Style Questionnaire
* Infant feeding history and food experience
* Toddler eating behaviors using the Child Eating Behavior Questionnaire for Toddlers
* Infant behaviors using the Infant Behavior Questionnaire-Revised (Garstein & Rothbart 2003 Inf Behav Dev)

ELIGIBILITY:
Inclusion Criteria:

* Term birth (at least 37 weeks gestation)
* Experience with complementary foods
* Previous exposure to nuts (butters, powders, or other nut ingredients)
* Caregiver at least 18 years of age and < 51 years of age
* Caregiver lives within 75 miles of the University of Colorado Anschutz Medical Campus
* Caregiver must feed the infant or toddler at least 50% of the time

Exclusion Criteria:

* Has a genetic disorder or developmental disability, as these conditions often result in feeding difficulties
* Has a reported illness or metabolic disorder (e.g., food allergy) that could affect food intake
* Was born prematurely (< 37 weeks gestation)
* Caregiver is less than 18 years of age
* Caregiver lives more than 75 miles from the University of Colorado Anschutz Medical Campus
* Caregiver does not read and speak English
* Caregiver has a food allergy

Ages: 7 Months to 24 Months | Sex: All
Age Groups: Child
Study Population: Infants and toddlers and their caregivers will be recruited for this study via:
  * printed advertisements placed in a number of community and healthcare venues and posted on online websites.
  * emails sent through the university
  * referrals from other participating caregivers
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in rate of infant acceptance of sweetened and unsweetened nutritional supplement | Baseline, Week 2
  Acceptance is measured at the conclusion of each offered bite using an adaptation of the Feeding Infants: Behavior and Facial Expression Coding System (FIBFECS) on a 4-point scale from 0-3 where 0 = refusal and 3 = early acceptance of food
Change in infant consumption of sweetened and unsweetened nutritional supplement | Baseline up to Week 2
  Consumption of each type of supplement will be measured in grams. The weight of the remainder of each supplement will be subtracted from the initial weight of the supplement prior to offering. The remainder of the supplements offered at home will be frozen and returned to the lab to be weighed.

SECONDARY OUTCOMES:
Baseline caregivers' perceived ratings of infant liking of sweetened and unsweetened supplements | Baseline
  After feeding each version of the supplement, the caregiver will be instructed to rate how much he/she thought his/her infant liked the supplement by placing a mark on a 100 mm visual analog scale (VAS) ranging from "dislikes extremely" to "likes extremely". The distance of the caregivers' marking on the 100mm line is measured from "dislikes extremely" in mm, with higher measurement values meaning caregivers perceive the infants like the supplement more.
Follow up caregivers' perceived ratings of infant liking of sweetened and unsweetened supplements | Visit two: change from baseline caregivers' perceived ratings at two weeks
  After feeding each version of the supplement, the caregiver will be instructed to rate how much he/she thought his/her infant liked the supplement by placing a mark on a 100 mm visual analog scale (VAS) ranging from "dislikes extremely" to "likes extremely". The distance of the caregivers' marking on the 100mm line is measured from "dislikes extremely" in mm, with higher measurement values meaning caregivers perceive the infants like the supplement more.
Baseline caregivers' perceived acceptability of the sweetened and unsweetened supplements | Baseline
  After feeding each version of the supplement, the caregiver will be instructed to rate how likely they would be to serve each supplement again by placing a mark on a 100 mm visual analog scale (VAS) ranging from "not at all likely" to "extremely likely". The distance of the caregivers' marking on the 100mm line is measured from "not at all likely" in mm, with higher measurement values meaning caregivers are more likely to serve the supplement again.
Follow up caregivers' perceived acceptability of the sweetened and unsweetened supplements | Visit two: change from baseline caregivers' acceptability ratings at two weeks
  After feeding each version of the supplement, the caregiver will be instructed to rate how likely they would be to serve each supplement again by placing a mark on a 100 mm visual analog scale (VAS) ranging from "not at all likely" to "extremely likely". The distance of the caregivers' marking on the 100mm line is measured from "not at all likely" in mm, with higher measurement values meaning caregivers are more likely to serve the supplement again.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Johnson, PhD, Principal Investigator — University of Colorado, Denver; Matthew Greenhawt, MD, Principal Investigator — University of Colorado, Denver; Jennifer O Fisher, PhD, Principal Investigator — Temple University; Kameron J Moding, PhD, Principal Investigator — Purdue University
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available upon request to the Principal Investigator (SL Johnson)

REFERENCES:
- [Background] Thompson AL, Mendez MA, Borja JB, Adair LS, Zimmer CR, Bentley ME. Development and validation of the Infant Feeding Style Questionnaire. Appetite. 2009 Oct;53(2):210-21. doi: 10.1016/j.appet.2009.06.010. Epub 2009 Jul 1. PMID 19576254
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Derived] Johnson SL, Shapiro ALB, Moding KJ, Flesher A, Davis K, Fisher JO. Infant and Toddler Consumption of Sweetened and Unsweetened Lipid Nutrient Supplements After 2-Week Home Repeated Exposures. J Nutr. 2021 Sep 4;151(9):2825-2834. doi: 10.1093/jn/nxab148. PMID 34036363